CLINICAL TRIAL: NCT01581632
Title: Assessment of Coronary Plaque Composition Using Near Infrared Spectroscopy During Inhibition of Lipoprotein-associated Phospholipase A2 (Lp-PLA2) Activity
Brief Title: Assessment of Coronary Plaque Composition
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Amir Lerman, Professor of Medicine, Mayo Clinic
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 09-007004
Record Dates: First submitted 2012-03-15; First posted 2012-04-20 (Estimated); Last update posted 2019-03-05 (Actual); Status verified 2017-11

CONDITIONS: Coronary Atherosclerosis; Endothelial Dysfunction; Coronary Small Vessel Disease
Keywords: atherosclerosis; endothelial dysfunction; coronary vasospasm
MeSH Terms: conditions — Coronary Artery Disease; Atherosclerosis; Coronary Vasospasm

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- LipiScan/LipiScan IVUS (Other): valuation of the coronary artery using near infrared spectroscopy using either a LipiScan catheter or a LipiScan/IVUS catheter following a clinically indicated coronary angiogram and endothelial function testing with a positive diagnosis of endothelial dysfunction. The procedure is repeated following 6 months of Lp-PLA2 inhibition.
  Interventions: Device: LipiScan/LipiScan IVUS

INTERVENTIONS:
Device: LipiScan/LipiScan IVUS — Evaluation of the coronary artery using near infrared spectroscopy using either a LipiScan catheter or a LipiScan/IVUS catheter following a clinically indicated coronary angiogram and endothelial function testing with a positive diagnosis of endothelial dysfunction. The procedure is repeated following 6 months of Lp-PLA2 inhibition.

SUMMARY:
The investigators' hypothesis is that local activation of the endogenous Lipoprotein-associated phospholipase A2 (Lp-PLA2) plays an integral role in early atherosclerosis, and contributes to the mechanism of coronary endothelial dysfunction and to the structural and mechanical properties that characterize plaque vulnerability. Thus, this study will characterize prospectively the correlation between the functional and structural vascular wall properties, and the activity of the Lp-PLA2 pathway.

DETAILED DESCRIPTION:
The present study will be a substudy of our National Institute of Health (NIH) funded and Institutional Review Board (IRB) approved (08-008161) protocol "Lp-PLA2 and Coronary Atherosclerosis in Humans" and (10-000044) "Lp-PLA2 and Coronary Atherosclerosis in Humans Aim III" in which the investigators are examining the impact of long-term inhibition of Lp-PLA2, with a specific novel inhibitor, on Lp-PLA2 activity and improvement in coronary endothelial function.

The substudy will allow the investigators to also examine the additional endpoint of lipid core content of atherosclerotic plaques and hence plaque vulnerability. Plaque lipid composition will be measured using the LipiScan or LipiScan IVUS catheter (InfraReDx Near Infrared Spectroscopy (NIRS) System with or without intravascular ultrasound (IVUS) capability) at baseline and again at 6 month following Lp-PLA2 inhibition.

The study will provide insight into the role of the endogenous Lp-PLA2 in early coronary atherosclerosis, a potential therapeutic target for early coronary atherosclerosis in humans.

ELIGIBILITY:
Inclusion Criteria:

* patients age > 18 years and < 85 years
* referred to our cardiac catheterization laboratory for coronary vasomotion testing- subsequently found to have coronary endothelial dysfunction.

Exclusion Criteria:

* heart failure ejection fraction <40%,
* unstable angina
* myocardial infarction or angioplasty within 6 months prior to entry into the study
* use of investigational agents within 1 month of entry into the study
* patients who require treatment with positive inotropic agents other than digoxin during the study
* patients with cerebrovascular accident within 6 months prior to entry the study
* significant endocrine, hepatic or renal, disorders, local or systemic infectious disease within 4 weeks prior to entry into study
* pregnancy or lactation
* mental instability

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2010-01; Primary Completion 2015-05 (Actual); Study Completion 2015-05 (Actual)

PRIMARY OUTCOMES:
Change from baseline of lipid plaque content measurement in the coronary artery | baseline and 6 month evaluation
  Following recruitment of the total study population and 6-months therapy with the Lp-PLA2 inhibitor, we will evaluate whether: 1. Plaque lipid content correlates with Lp-PLA2 levels and endothelial function 2. Lp-PLA2 inhibition reduced coronary plaque lipid content

CONTACTS AND LOCATIONS:
Overall Officials: Amir Lerman, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials